CLINICAL TRIAL: NCT04062032
Title: Pilot Studies Assessing the Metabolomic and Inflammatory Effects of Oral Aspirin (ASA) in Human Subjects at Risk for Melanoma
Brief Title: Metabolomic and Inflammatory Effects of Oral Aspirin (ASA) in Subjects at Risk for Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCI94424 Pilot
Record Dates: First submitted 2019-08-13; First posted 2019-08-20 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASA 81 mg daily (Experimental): Participants will be given ASA 81 mg orally once daily for a total of 7 days
  Interventions: Drug: Aspirin 81 mg
- ASA 325 mg daily (Experimental): Participants will be given ASA 325 mg orally once daily for a total of 7 days.
  Interventions: Drug: Aspirin 325mg

INTERVENTIONS:
Drug: Aspirin 81 mg — ASA 81mg taken daily
  Other Names: ASA
  Arms: ASA 81 mg daily
Drug: Aspirin 325mg — ASA 325mg taken daily
  Other Names: ASA
  Arms: ASA 325 mg daily

SUMMARY:
This is an open label phase II pilot study assessing the metabolomic and inflammatory effects of oral aspirin (ASA) in human subjects at risk for melanoma.

DETAILED DESCRIPTION:
Primary Objectives

I. Open label trial in 60 patients to assess the capacity of either of one daily dose (81, 325 mg) of sub-chronic ASA administration to increase the plasma and nevus ASA metabolites such as: salicylate, salicylurate, gentisic acid, and salicyl acyl glucuronide.

II. Open label trial in 60 patients to assess the capacity of sub-chronic daily ASA (81, 325 mg) administration to reduce levels of prostaglandin E2 (PGE2) in plasma and nevi.

Secondary Objectives

I. Determine whether ASA increases AMP-activated protein kinase (AMPK) activation in nevi.

II. Determine whether ASA affects whole blood leukocytes or leukocyte subsets in plasma.

III. Determine whether ASA affects inflammatory cytokines in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 2 nevi (each >5 mm diameter) not clinically suspicious for melanoma that can be biopsied.
* Must be older than age 18.
* Must be able to receive informed consent and sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* The patient is a minor, under age 18.
* The patient cannot speak / understand English or Spanish.
* The patient is pregnant or breastfeeding.
* The patient is a prisoner, critically or mentally ill, or otherwise incapacitated or considered vulnerable.
* The patient has history of allergic reaction to ASA.
* The patient has history of severe asthma.
* The patient has been taking ASA or any NSAID in the past 2 weeks.
* The patient has been taking a blood thinner in the past 2 weeks.
* The patient has history of bleeding disorder.
* The patient has history of peptic ulcer disease.
* The patient has had recent intense UV exposure in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Change in concentration of ASA metabolites (salicylate and salicylurate) in plasma after ASA ingestion | Change from baseline to day 7
  Concentration (ng/mL) of pre-treatment ASA metabolites (salicylate and salicylurate) in plasma will be compared to the concentration of ASA metabolites at day 7
Change in concentration of ASA metabolites in nevus tissue after ASA ingestion | Change from baseline to day 7
  Pre-treatment ASA metabolites in tissue will be compared to ASA metabolites at day 7
Change in concentration of prostaglandin E2 (PGE2) in plasma after ASA ingestion | Change from baseline to day 7
  Baseline PGE2 levels in plasma specimens will be compared to PGE2 levels at day 7.
Change in concentration of prostaglandin E2 (PGE2) in nevus tissue after ASA ingestion | Change from baseline to day 7
  Baseline PGE2 levels in tissue specimens will be compared to PGE2 levels at day 7.

SECONDARY OUTCOMES:
Change in AMP-activated protein kinase (AMPK) activation in nevi after ASA ingestion | Change from baseline to day 7
  Quantitative densitometry analysis using Western blots will be performed on tissue collected at baseline and at day 7 to compare activation of AMP-activated protein kinase (AMPK).
Change in concentration of leukocytes in peripheral blood after ASA ingestion | Change from baseline to day 7
  Whole blood will be taken at baseline and at day 7 to compare concentration of leukocytes

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Grossman, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States